CLINICAL TRIAL: NCT00154869
Title: An Open Label, Comparative, Multi-Center Study, to Evaluate the Efficacy and Safety of Peginterferon Alfa-2a Plus Ribavirin in the Treatment of Patients With Chronic Hepatitis C/Hepatitis B Co-Infection and Chronic Hepatitis C
Brief Title: Peginterferon Alfa-2a Plus Ribavirin for Chronic Hepatitis C/Hepatitis B Co-Infection and Chronic Hepatitis C
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 921003; ML17862
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-08-13 (Estimated); Status verified 2005-08

CONDITIONS: Hepatitis B, Chronic; Hepatitis C, Chronic
Keywords: Patients with dual chronic hepatitis B and C
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

INTERVENTIONS:
Drug: Peginterferon Alfa-2a plus Ribavirin

SUMMARY:
The investigators' pilot study indicates that hepatitis C virus (HCV)- and hepatitis B virus (HBV)-coinfected patients with predominantly active hepatitis C and those with predominantly active hepatitis B may need different anti-viral regimens. Since in the majority of these coinfected patients the hepatitis activity is more likely due to HCV than to HBV, the optimal therapeutic regimen for HCV- and HBV-coinfected patients with predominantly active hepatitis C will first be investigated. The combination therapy using pegylated interferons (IFNs) such as PEG-IFN alfa-2a has been shown to have a superior efficacy than that using conventional IFN in the treatment of monoinfected chronic hepatitis C. This new combination therapy might also further enhance the treatment efficacy in HCV- and HBV- coinfected patients. The investigators therefore propose to initiate a trial comparing the efficacy of pegylated IFN plus ribavirin (RBV) in dual chronic hepatitis B and C versus that in chronic hepatitis C only, for both HCV genotype 1 and 2/3 patients. The efficacy using a 24-week combination therapy in the sustained clearance of serum HCV RNA is equivalent to that using a 48-week combination therapy in patients with HCV genotype non-1 [Hadziyannis et al, EASL 2002]. A 48-week course of pegylated IFN and RBV combination therapy, in contrast, has been shown to yield a better efficacy in the sustained clearance of serum HCV RNA in patients with HCV genotype 1 than a 24-week combination therapy in western countries [Hadziyannis et al, EASL 2002; Poynard et al, 1998]. The primary objective of the current proposal is to investigate and compare the efficacy of combination therapy using pegylated IFN plus RBV on the clearance of serum HCV RNA in both dually infected patients with a dominant HCV infection and HCV monoinfected patients. Therefore, in this proposal, the treatment duration will be 24 weeks for HCV genotype 2/3 in patients with dual chronic hepatitis C and B and in patients with monoinfected HCV, and will be 48 weeks for HCV genotype 1 in patients with dual chronic hepatitis C and B and in patients with monoinfected HCV.

DETAILED DESCRIPTION:
Around the world, the majority of hepatitis C patients suffer a monoinfected chronic HCV infection. Current regimen on this group of patients received much attention and resulted in rapid advances [McHutchison et al, 1998]. However, there are certain understudied populations with chronic hepatitis C [Strader DB, 2002]. One important group of them is the patients co-infected by HBV. In hepatitis B or C endemic areas, the number of subjects with dual infections of both hepatitis C and B is substantial [Chen et al, 1990; Tsai et al, 1994; Liaw 1995; Pramoolsinsap et al, 1999]. For example, in Taiwan, anti-HCV was present in 11% of patients with HBV-related chronic liver diseases [Chen et al 1990; Liaw 1995], and HBsAg positive rate was 12% in anti-HCV-positive patients [Tsai et al, 1994]. In Italy, the prevalence of anti-HCV positivity can be as high as 40% in patients with chronic active hepatitis B in some cities [Sagnelli et al, 1997]. Such co-infected patients are rarely encountered in the developed countries, except in intravenous drug users, hemophiliacs or those receiving hemodialysis. Alarmingly, the HCV- and HBV- coinfected patients have been shown to carry a greater risk (1.5~5 folds) of developing LC or HCC than those with HCV or HBV infection only [Liaw 1995; Donato et al, 1998; Yang et al, 2002; Sun et al, 2003]. Therefore, the HBV and HCV dually infected patients also need active treatments. Unfortunately, current therapeutic targets and ongoing protocols of clinical trials recruit patients with HCV infection only and invariably exclude those co-infected with HBV. Thus, it is warranted to address this important issue and an effective treatment for these hepatitis C and B dually infected patients is desperately needed.

Sporadic studies showed that IFN alone was not effective in clearing HCV or HBV in patients dually infected with hepatitis B and C [Liaw 1995; Liaw et al, 1997; Weltman et al, 1995; Mazzella et al, 1999; Guptan et al, 1999]. A recent study reported that dose augmentation of IFN to 9 MU thrice weekly for 6 months could clear HCV in 31% of the patients [Villa et al, 2001]. Apparently, the efficacy was still not adequate. Because combining IFN with RBV has been shown to yield much better results in the treatment of chronic hepatitis C than IFN alone [Poynard et al, 1995; Davis et al, 1998; Reichard et al, 1998; McHutchison et al, 1998; Lai et al, 1996; Liaw et al, 1997; Schalm et al, 1999], the combination therapy might also be more effective in treating dual hepatitis B and C patients. To test this, we conducted a pilot study using conventional IFN alfa plus ribavirin to treat 24 patients coinfected with HCV and HBV. The 24-week combination regimen with IFN and ribavirin cleared HCV in 43% (9/21) of the patients dually infected with hepatitis B and C. The result was comparable to that in patients with monoinfected chronic hepatitis C. Normalization of serum ALT was obtained in 38% of the patients 24 weeks after the end of the treatment. In addition, we found that although the end-of-treatment clearance rate of HCV RNA was comparable between patients infected with genotype 1b and those with genotype 2a or 2b, the clearance of HCV RNA sustained much less commonly in those infected by HCV genotype 1b (21% vs. 86%, P<0.05). Actually, two recent studies from southern Taiwan also demonstrated that the efficacy of combination therapy using interferon plus ribavirin on the clearance of serum HCV RNA was comparable between HBV and HCV coinfected patients versus HCV monoinfected patients [Wang et al., 2003; Yu et al., 2003]. Based on these findings, we suggested that comparable efficacy of combination therapy using interferon plus ribavirin on the clearance of serum HCV RNA can be achieved in patients with HBV and HCV coinfected patients versus HCV monoinfected patients. Nevertheless, a more effective regimen is still needed for those dually infected patients, particularly for those with HCV genotype 1.

In our pilot study, we treated 24 patients coinfected with HCV and HBV as a single group. The majority of these patients had detectable hepatitis C viremia, but were anti-HBe positive and with a lower serum HBV titer. Therefore, hepatitic activity was more likely due to HCV than to HBV. Nevertheless, a few patients were HBeAg positive and had a higher serum HBV titer (>105 copies/mL) but with a low or undetectable serum HCV RNA. In them, the hepatitis was likely due to active hepatitis B. Importantly; none of the dually infected patients with predominantly active hepatitis B had biochemical and HCV virologic response both at the end of combination therapy and at 24 weeks post-treatment follow-up. These two groups of patients may need different anti-viral regimens according to the major offending virus in the liver. To treat dual hepatitis C and B patients with dominantly active hepatitis C, we may use IFN (conventional or pegylated form) and RBV, and the treatment schedule may be extended to one year to enhance the efficacy for those with HCV genotype 1. However, to treat dually infected patients with a dominant HBV infection, the treatment strategy may be different.

Our pilot study indicates that HCV- and HBV-coinfected patients with predominantly active hepatitis C and those with predominantly active hepatitis B may need different anti-viral regimens. Since in the majority of these coinfected patients the hepatitis activity is more likely due to HCV than to HBV, the optimal therapeutic regimen for HCV- and HBV-coinfected patients with predominantly active hepatitis C will first be investigated. The combination therapy using pegylated IFNs such as PEG-IFN alfa-2a has been shown to have a superior efficacy than that using conventional IFN in the treatment of monoinfected chronic hepatitis C. This new combination therapy might also further enhance the treatment efficacy in HCV- and HBV- coinfected patients. We therefore propose to initiate a trial comparing the efficacy of pegylated IFN plus RBV in dual chronic hepatitis B and C vs. that in chronic hepatitis C only, for both HCV genotype 1 and 2/3 patients. The efficacy using a 24-week combination therapy in the sustained clearance of serum HCV RNA is equivalent to that using a 48-week combination therapy in patients with HCV genotype non-1 [Hadziyannis et al, EASL 2002]. A 48-week course of pegylated IFN and RBV combination therapy, in contrast, has been shown to yield a better efficacy in the sustained clearance of serum HCV RNA in patients with HCV genotype 1 than a 24-week combination therapy in western countries [Hadziyannis et al, EASL 2002; Poynard et al, 1998]. The primary objective of the current proposal is to investigate and compare the efficacy of combination therapy using pegylated IFN plus RBV on the clearance of serum HCV RNA in both dually infected patients with a dominant HCV infection and HCV monoinfected patients. Therefore, in this proposal, the treatment duration will be 24 weeks for HCV genotype 2/3 in patients with dual chronic hepatitis C and B and in patients with monoinfected HCV, and will be 48 weeks for HCV genotype 1 in patients with dual chronic hepatitis C and B and in patients with monoinfected HCV.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients >= 18 years of age will be recruited.
* Patients with dual chronic hepatitis C and B must be positive for both anti-HCV and HBsAg for more than 6 months and HCV RNA quantifiable at 600 IU/mL (by the COBAS AMPLICOR HCV MONITOR® Test version 2.0).
* Patients must not be positive for HBeAg.
* Patients with monoinfected chronic hepatitis C must be positive for anti-HCV for more than 6 months and HCV RNA quantifiable at 600 IU/mL (by the COBAS AMPLICOR HCV MONITOR® Test version 2.0). Patients must not be positive for HBsAg.

All patients must:

* Be treatment naïve for the hepatitis disease or have had treatment failure to previous interferon monotherapy or treatment failure to previous lamivudine therapy.
* Present with elevated serum ALT levels at least 1.5 times the upper limit of normal, documented on two occasions (at least one month apart), within six months prior to enrollment
* Present with liver biopsy findings compatible with the diagnosis of chronic liver disease (the liver biopsy needs to be taken within 52 weeks prior to the first dose of study drug)
* Have adequate liver reserve (defined as equal to or better than Child-Pugh Class A)
* Present with WBC 3500/mm3, ANC 1500/mm3, and platelets 90,000/mm3

Exclusion Criteria:

* Be drug addicts or have any history or histological evidence of alcohol abuse, or currently receive prescriptions that may cause hepatotoxicity
* Present with hemoglobin <12.0 gm/dl for females and <13.0 gm/dl for males
* Signs or symptoms of hepatocellular carcinoma
* Any investigational drug ? 6 weeks prior to the first dose of study drug
* Have renal insufficiency (serum creatinine concentration >1.5 x upper limit of normal at screening; upper limit depending on lab at each site)
* Patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled if, in the judgment of the investigator, an acute decrease in hemoglobin by up to 4 g/dL (40 g/L) (as may be seen with ribavirin therapy) would not be well-tolerated.
* Have serological evidence of autoimmune chronic liver disease (e.g. antinuclear antibody titers > 1:320, and/or smooth muscle antibody titers > 1:160)
* History of major organ transplantation with an existing functional graft
* History or other evidence of severe illness, malignancy or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* Thyroid dysfunction not adequately controlled (TSH and T4 levels out of normal range)
* Evidence of severe retinopathy (e.g., CMV retinitis, macular degeneration) or clinically relevant ophthalmological disorder due to diabetes mellitus or hypertension
* Have been exposed to hepatotoxic substances which might be the cause of hepatitis
* Be pregnant, lactating or not practicing two adequate forms of birth control, such as oral contraceptives or intrauterine devices
* Be seropositive for anti-HIV or anti-delta or anti-HAV IgM Ab
* History of severe psychiatric disease, especially depression, characterized by a suicide attempt, hospitalization for psychiatric disease, or a period of disability as a result of psychiatric disease
* Have AFP (alpha-fetoprotein) greater than 20 ng/ml; in case of elevated AFP, abdomen ultrasonography is required to exclude the possibility of HCC.
* History of severe cardiac disease (e.g., NYHA Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina or other significant cardiovascular diseases).
* Have a history of asthma (see above) or drug allergy which may lead to the hypersensitivity to ribavirin
* Male partners of women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2004-06; Study Completion 2007-08

PRIMARY OUTCOMES:
To demonstrate the efficacy of peginterferon alfa-2a (PEG-IFN alfa-2a) (Pegasys®) plus ribavirin (RBV) for sustained virological response (SVR) in HBV-coinfected versus monoinfected chronic hepatitis C (CHC) patients

SECONDARY OUTCOMES:
To demonstrate the efficacy of peginterferon alfa-2a (PEG-IFN alfa-2a) (Pegasys®) plus ribavirin (RBV) on the reduction of HCV viremia after 24 and 48 weeks of treatment (depending on genotype) in coinfected versus monoinfected CHC patients
To demonstrate the efficacy of PEG-IFN alfa-2a plus RBV in dual chronic hepatitis C and B on:
1) the biochemical response rate
2) the score of histologic change
3) serum HBV DNA disappearance
4) HBsAg disappearance
5) combined response of HBV DNA disappearance and normalization of ALT
6) end of treatment virological response
To assess the influence of serum HBV load on the clearance of serum HCV RNA, the loss of serum HBV DNA, and normalization of serum ALT
To assess the influence of HBV genotype on the clearance of serum HCV RNA, the loss of serum HBV DNA, and normalization of serum ALT
To assess the safety profile of the PEG-IFN alfa-2a plus RBV combination therapy in dual chronic hepatitis C and B

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jer Chen, M.D.; Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Internal Medicine, Taipei, Taiwan